CLINICAL TRIAL: NCT07089524
Title: A Comparative Study Between Neutrophil/Lymphocyte Ratio and Lactate/Albumin Ratio as Predictive Inflammatory Markers for Sepsis in Patients With Lower Respiratory Tract Infection in ICU
Brief Title: A Comparative Study Between Neutrophil/Lymphocyte Ratio and Lactate/Albumin Ratio as Predictive Inflammatory Markers for Sepsis
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD210/2024
Record Dates: First submitted 2025-04-04; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational group (160 patients ): Data collection: (upon admission to ICU)
  All the study subjects will be submitted to:
  I) Careful clinical evaluation including:
  * Demographics.
  * Comorbid conditions.
  * Medication usage (including intravenous fluids and vasoactive medications).
  * Vital signs .
  * Mental status (Glasgow Coma Score)
  * SOFA (Sequential Organ Failure Assessment) score.
  * Duration of antibiotics treatment.
  II) Laboratory Investigations including:
  * Complete blood picture (CBC): including Neutrophils and Lymphocytes count.
  * Serum albumin and serum lactate.
  * Prothrombin time and concentrations.
  * Liver function tests (LFTs), serum creatinine and urea.
  * Electrolytes, arterial blood gases.
  * Highly sensitive C -reactive protein (Hs CRP).
  III) Microbiological investigations:
  Various body fluid cultures, including sputum, blood, and urine will be obtained to identify source of sepsis.
  All investigations will be done at Ain Shams University, central lab unit.

SUMMARY:
Aim of this study is to predict the prognostic values of Neutrophil/ Lymphocyte ratio and Lactate/Albumin ratio in the outcome of patients with sepsis and septic shock with lower respiratory tract infection, also to compare between them regarding sensitivity and specificity.

DETAILED DESCRIPTION:
Lower respiratory tract infection (LRTI) is one of the most common infectious diseases that lead to admission of patients to ICU. It includes a wide range of respiratory infections; such as pneumonia, bronchitis, empyema and lung abscess. Furthermore, it is associated with considerable morbidity and mortality. Because delay in the ICU admission of patients with LRTI has been shown to be associated with increased mortality, it can be helpful to predict the mortality of LRTI patients in hospitals.

Sepsis is a life-threatening medical emergency induced by uncontrolled systemic inflammatory response of the host to infection. Without an early and aggressive management, sepsis can rapidly lead to organ failure, tissue hypoperfusion, and death. Bacterial infections cause most cases of sepsis, but it can also be a result of other infections; such as viral, fungal or parasitic infections. Sepsis-3 definitions for sepsis management were established in 2016 according to the Surviving Sepsis Campaign guidelines. They define sepsis as "a life-threatening organ dysfunction caused by a dysregulated host response to infection", and septic shock as "a subset of sepsis in which underling circulatory and cellular/metabolic abnormalities are profound enough to substantially increase mortality".

According to Sepsis-3 criteria, sepsis and septic shock are currently diagnosed as follows: sepsis-suspected or documented infection plus SOFA (Sequential Organ Failure Assessment) score ≥2; septic shock-sepsis plus vasopressor therapy needed to maintain mean arterial pressure (MAP) ≥65 mmHg plus lactate ≥2 mmol/L (18 mg/L) despite adequate fluid resuscitation. However these diagnosis criteria, the early evaluation of sepsis severity and prognosis is still imprecise and significant research is being performed to address this issue.

The neutrophil/lymphocyte ratio (NLR) was studied in order to provide an easier way to diagnose sepsis. This ratio can be calculated both from the absolute number of neutrophils and lymphocytes, and from their relative number. The importance of this report derives from the fact that physiological stress causes an increase in the number of neutrophils and a decrease in the number of lymphocytes. Sepsis stimulates lymphocyte apoptosis, so this ratio is increased in these cases. Septic shock causes a dramatic decrease in lymphocyte count, so the NLR ratio increases significantly.

Increased lactate production is a prognostic marker of generalized hypoxia in distributive shock. Previous studies have reported that lactate levels are a dependable parameter in diagnosis, therapeutic evaluation, and prognosis in circulatory shock. Increased lactate levels are used worldwide for early diagnosis, management, and in risk stratification of patients with septic shock .

Albumin is a negative acute-phase protein, and its levels can reflect the magnitude of inflammation. In critically ill patients, the degree of hypoalbuminemia thus represents the severity of the inflammatory response. Consequently, it may be a prognostic biomarker in patients with sepsis .

Although lactate and albumin values independently predict mortality, the ratio of lactate to albumin (L/A ratio) is superior as a predictor to lactate or albumin alone. This result has been recorded in studies conducted in recent years .

ELIGIBILITY:
Inclusion Criteria:

* Adults with lower respiratory tract infection
* Confirmed septic patients (under the third international consensus definitions of sepsis and septic shock),
* Admitted to intensive care unit.
* Age (18-80) years.
* Both genders.

Exclusion Criteria:

* Age: < 18 years old, > 80 years old
* Patient refusal.
* Pregnancy.
* Malignancy.
* Pathology that could affect serum albumin concentrations prior to ICU admission as Malnutrition
* Nephrotic syndrome
* Liver Cirrhosis
* Intestinal resection surgeries

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with lower respiratory tract infection confirmed septic patients admitted to Ain Shams University Hospitals ICU
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Detect the mortality due to sepsis with lower respiratory tract infection | From date of randomization until the date of death during the study period ( 12-18 months)
  Detect the mortality due to sepsis and septic shock in patients with lower respiratory tract infection in ICU
The prognostic values of Neutrophil/Lymphocyte ratio and Lactate/Albumin ratio in Sepsis | From date of randomization until the date of discharge from the ICU or death during the study period ( 12-18 months )
  predict the prognostic values of Neutrophil/Lymphocyte ratio and Lactate/Albumin ratio in the outcome of septic patients with lower respiratory tract infection in ICU

SECONDARY OUTCOMES:
The duration of intensive care unit stay | From date of randomization until the date of discharge from the ICU or death during the study period ( 12-18 months )
  The duration of intensive care unit stay in days from admission to ICU until discharge or death during the period of the study (12-18 months)
The requirement for vasoactive medications | From date of randomization until the date of discharge from the ICU or death during the study period ( 12-18 months )
  The requirement for vasoactive medications regarding the doses in microgram per kilogram per minute and the duration in days
Mechanical ventilatory support and renal replacement therapy | From date of randomization until the date of discharge from the ICU or death during the study period ( 12-18 months )
  The need of mechanical ventilatory support and the need of renal replacement therapy and its duration in days

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No